CLINICAL TRIAL: NCT06216431
Title: Investigation of Respiratory System, Musculoskeletal System, Physical Activity Level and Quality of Life in Different Types of Office Workers.
Brief Title: Respiratory and Physical Outcomes in Different Types of Office Workers
Status: Active, not recruiting | Type: Observational
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Gulsah Bargi, Principal Investigator, Izmir Democracy University
Other Study IDs: Different Office Workers
Record Dates: First submitted 2023-12-29; First posted 2024-01-22 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Work-related Illness
Keywords: office workers; call center operators; musculoskeletal discomfort; dyspnea; posture; thoracic mobility
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Emergency call center workers: This group will consist of individuals working as operators at Izmir 112 Emergency Call Center.
  Interventions: Other: Physical Evaluations of individuals
- Office workers: This group will consist of office workers who work actively at a desk.
  Interventions: Other: Physical Evaluations of individuals

INTERVENTIONS:
Other: Physical Evaluations of individuals — Participants will be evaluated on posture, chest mobility, cough strength, flexibility, hand grip strength and pinch strength. They will be asked to answer the Modified Medical Research Council Scale, Cornell Musculoskeletal Disorders Questionnaire, International Physical Activity Questionnaire Short Form and Short Form -36. The data to be obtained from all these evaluations are planned to be collected face to face from the participants at once and within a maximum of 1 hour.

SUMMARY:
There are no studies in the literature reporting the posture, chest mobility, dyspnea, flexibility, quality of life and physical activity levels of emergency call center employees. The aims of this observational study are; 1) to evaluate posture, chest mobility, strength, dyspnea, flexibility, musculoskeletal disorders, physical activity and quality of life in emergency call center workers and office workers, 2) to reveal the relationships between these parameters of both research groups and 3) The aim is to compare these measurement parameters in emergency call center workers and office workers.

DETAILED DESCRIPTION:
Over time, there has been an increase in the number of office workers and the use of computers. Working in a static position for long working hours and improper working postures can lead to loss of flexibility in the muscles, decrease in thoracic mobility, pain in the musculoskeletal system and deterioration of ideal posture. Emergency call center employees work long hours, in shifts that require serious attention, where stress is intense and the circadian rhythm is disrupted. There is no study in the literature that evaluates the posture, chest mobility, dyspnea, flexibility and physical activity levels of emergency call center employees. Therefore, the aim of our study is; It is a comparative evaluation of posture, chest mobility, cough strength, dyspnea flexibility, musculoskeletal disorders, physical activity level and quality of life in emergency call center operators and desk workers.

ELIGIBILITY:
Inclusion Criteria for Emergency Call Center Workers

* Being an operator at Izmir 112 Emergency Call Center
* Being 18 years or older
* Volunteering to participate in the study
* Being able to understand and answer surveys

Inclusion Criteria for Office Workers

* Being actively working at a desk
* Being 18 years or older
* Volunteering to participate in the study
* Being able to understand and answer surveys

Exclusion Criteria:

* Have any history of acute/chronic infection, physical or mental disability/disease and/or cognitive impairment that would prevent measurement.
* Being pregnant
* Being able to exercise regularly

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: At least 27 individuals will be included in the emergency call center workers group and at least 25 individuals will be included in the office workers group.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Handgrip strength | up to 5 minutes
  Hand grip strength will be measured using the Jamar hand dynamometer.

SECONDARY OUTCOMES:
Thoracic mobility | up to 5 minutes
  Individuals will be asked to sit in an upright sitting position with their arms slightly open, and their chest circumference will be measured with a tape measure at three different levels (axillary, epigastric, subcostal) at rest, deep breathing (maximum inspiration) and deep exhalation (maximum expiration). The difference between measurements will be recorded in centimeters.
Cough strength | up to 2-3 minutes
  Cough strength will be evaluated using a PEFmeter.
Dyspnea | up to 1 minute
  Dyspnea will be assessed using the Modified Medical Research Council (MMRC) Scale. This scale is a five-item scale based on various physical activities that cause a feeling of shortness of breath (dyspnea). As the score an individual gets from the scale increases, the perception of shortness of breath also increases.
Posture | up to 5 minutes
  Posture will be evaluated with sensorless posture analysis software based on the artificial intelligence concept created by Fizyosoft and Becure.
Musculoskeletal pain | up to 5 minutes
  Musculoskeletal pain will be assessed using the Turkish version of the Cornell Musculoskeletal Disorders Questionnaire. The score is obtained by multiplying the weighted scores corresponding to the individual's answer. The scores obtained for each region range between 0 and 90, and higher scores indicate higher levels of pain disorder.
Flexibility | up to 5 minutes
  Flexibility will be evaluated with sit-reach test, pectoral shortness tests, and shoulder adductor and internal rotator shortness tests.
Pinch strength | up to 5 minutes
  Pinch strength will be evaluated using a hydraulic pinch dynamometer.
Physical activity level | up to 2 minutes
  Physical activity level will be assessed using the Turkish version of the International Physical Activity Questionnaire Short Form."MET-min/week" scores were obtained by multiplying the minutes, days, and MET (which is set by convention at 3.5 milliliter of oxygen per kilogram per minute) values of each activity. According to these scores, individuals were classified as inactive, minimally active, and sufficiently active.
Health-related quality of life | up to 5 minutes
  Quality of life will be assessed using the SF-36. It consists of eight subscales including physical function, role limitations due to physical health and emotional problems, vitality, emotional well-being, social function, bodily pain, and general health. Each subscale is scored between 0 (poorer health) and 100 (better health).

CONTACTS AND LOCATIONS:
Overall Officials: GÜLŞAH BARĞI, Assoc.Dr., Study Director — Izmir Democracy University; BERFİN KİŞİN, MSc, Principal Investigator — Izmir Emergency Call Center; ÖZLEM ÇİNAR ÖZDEMİR, Assoc.Dr., Principal Investigator — Izmir Democracy University
Locations (1):
- Izmir Democracy University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clemes SA, O'Connell SE, Edwardson CL. Office workers' objectively measured sedentary behavior and physical activity during and outside working hours. J Occup Environ Med. 2014 Mar;56(3):298-303. doi: 10.1097/JOM.0000000000000101. PMID 24603203
- [Background] Heneghan NR, Baker G, Thomas K, Falla D, Rushton A. What is the effect of prolonged sitting and physical activity on thoracic spine mobility? An observational study of young adults in a UK university setting. BMJ Open. 2018 May 5;8(5):e019371. doi: 10.1136/bmjopen-2017-019371. PMID 29730619
- [Background] Janwantanakul P, Pensri P, Jiamjarasrangsri V, Sinsongsook T. Prevalence of self-reported musculoskeletal symptoms among office workers. Occup Med (Lond). 2008 Sep;58(6):436-8. doi: 10.1093/occmed/kqn072. Epub 2008 Jun 10. PMID 18544589
- [Background] Rostamzadeh S, Saremi M, Fereshteh T. Maximum handgrip strength as a function of type of work and hand-forearm dimensions. Work. 2020;65(3):679-687. doi: 10.3233/WOR-203100. PMID 32116266